CLINICAL TRIAL: NCT06890195
Title: Effect of Dialysate Cooling Versus Sodium Profiling in Management of Intradialytic Hypotension Among Chronic Hemodialysis Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Samir Abbas, Rsidant doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: cooling VS sodium profilingIDH
Record Dates: First submitted 2025-03-17; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Intradialytic Hypotension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Active Comparator): dialysate cooling group: patients will be subjected to individualized cool dialysate (dialysate temperature 0.5 °C lower than core body temperature)
  Interventions: Procedure: dialysate cooling
- Group B (Placebo Comparator): sodium profiling group: patients will be subjected to standard dialysate temperature (dialysate temperature of 37 °C).
  Interventions: Procedure: standard dialysate temperature

INTERVENTIONS:
Procedure: dialysate cooling — patients will be subjected to individualized cool dialysate (dialysate temperature 0.5 °C lower than core body temperature)
  Arms: Group A
Procedure: standard dialysate temperature — patients will be subjected to standard dialysate temperature (dialysate temperature of 37 °C).
  Arms: Group B

SUMMARY:
Chronic kidney disease (CKD) is a worldwide public health issue. Dialysis patients have a tenfold greater relative risk of cardiovascular death than the general population.

Dialysate cooling prevents intradialytic hypotension (IDH). This is achieved by inducing vasoconstriction and activating the sympathetic nervous and therefore improving hemodynamic stability .

Intradialytic hypotension (IDH) is a common complication of HD. There is no consensus on the definition of IDH, but (IDH) is commonly defined as a drop in blood pressure during dialysis procedure and/ or hypotensive symptoms such as dizziness, weakness, nausea, cramps, blurred vision, and fatigue .

The pathophysiology of IDH is diverse. It could be the result of an inadequate cardiovascular response to the reduction in blood volume that occurs when the ultrafiltration volume is large . One process may involve an imbalance between a reduced effective circulating volume and the compensatory plasma refilling mechanism, wherein fluid from the interstitial and intracellular space is translocated into the intravascular compartment .

Cold dialysis reduces HD-induced brain damage by protecting the cerebral vascular beds from harmful perfusion . In the heart, long- term cold dialysis improved resting ejection fraction and reduced left ventricular mass and end-diastolic volumes while preserving aortic distensibility, decreasing the risk for future cardiovascular events

. Risk factors associated with IDH include old age, female gender, Hispanic ethnicity, long dialysis vintage, high intradialytic weight gain, high dialysis dose, anemia, diabetes, low pre-dialysis BP, high osmolarity, and high body mass index .

It can be applied universally and reduce the need for nursing involvement . Further, no additional cost is needed to conduct fixed reduction of dialysate temperature. While there are various methods of reducing dialysate temperature, optimal temperature or methods of temperature reduction to prevent IDH remain uncertain

To study the effect of dialysate cooling (0.5- 1 C lower than pre- dialysis core body temperature) Vs traditional sodium profiling on:

1. Reduction the episodes of IDH .
2. Net dry weight achievements.
3. Post dialysis fatigue.

ELIGIBILITY:
Inclusion Criteria:

* • Patients age 18-70 years old.

  * Maintained on HD for not less than 6 months
  * Documented episodes of IDH

Exclusion Criteria:

* • Severly anemic patients (Hb<7 g/dl)

  * Patients taking more than 3 antihypertensive (on days other than dialysis day).
  * Patients with documented IHD.
  * Patients on midodraine therapy prior dialysis session.
  * patient refusal, incompliance or ineffective dialysis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
number in IDH episodes | 6 week
  compare the total number in IDH episodes and Frequency of hypotensive symptoms between two group